CLINICAL TRIAL: NCT01049399
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study Evaluating the Safety, Tolerability, and Efficacy of Two Different Oral Doses of NP031112, a GSK-3 Inhibitor, Versus Placebo in the Treatment of Patients With Mild-to-Moderate Progressive Supranuclear Palsy
Brief Title: Safety, Tolerability, and Efficacy of Two Different Oral Doses of NP031112 Versus Placebo in the Treatment of Patients With Mild-to-Moderate Progressive Supranuclear Palsy
Acronym: Tauros
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noscira SA (Industry)
Collaborators: i3 Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP031112-08B02
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): once daily administration of powder for oral suspension.
  Interventions: Drug: placebo
- NP031112 800 mg (Experimental): Group dosed with 800 mg once daily for 52 weeks
  Interventions: Drug: tideglusib
- NP031112 600 mg (Experimental): Group treated with 600 mg once daily for 52 weeks
  Interventions: Drug: tideglusib

INTERVENTIONS:
Drug: tideglusib — 800 mg of tideglusib as a powder for oral suspension once daily in fasting conditions for 52 weeks
  Other Names: NP031112
  Arms: NP031112 800 mg
Drug: tideglusib — 600 mg of tideglusib as a powder for oral suspension, administered once daily in fasting conditions for 52 weeks
  Other Names: NP031112
  Arms: NP031112 600 mg
Drug: placebo — powder for oral suspension administered once daily in fasting conditions for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine wether NP031112 is safe and effective in the treatment of mild to moderate Progressive Supranuclear Palsy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with diagnosis of possible or probable PSP according to clinical criteria of National Institute of Neurologic Diseases and Stroke - the Society for PSP (Appendix 1).
2. Age of 40 to 85 years (patients over 85 years could be included after previous assessment by Investigator and approved by sponsor).
3. Brain magnetic resonance imaging (MRI) study within 24 months before Baseline visit excluding other potential causes of parkinsonism, especially cerebrovascular lesions and space occupying lesions.
4. Mild-to-moderate stage of disease severity according to score of 1 to 4 in Golbe Staging System.(Appendix 2)
5. Female patients must be surgically sterilized; at least 1 year postmenopausal (confirmed by follicle-stimulating hormone [FSH] >20 international units [IUs]); using adequate birth control (implants, injectables, combined oral contraceptives, intrauterine contraceptive device, total sexual abstinence during the study or vasectomised partner). Male patients must be willing to use barrier contraception (condom) during the study and for 6 months after last treatment administration.

   In European arms of study female patients must be without childbearing potential.
6. Caregiver (or dedicated nurse) living in same household or interacting with patient for >4 hours every day able to assure correct preparation and administration of study drug.
7. Patients living at home or in retirement home not requiring continuous nursing care.
8. General health status acceptable for participation in 64-week clinical trial.
9. Ability to swallow 100 mL of water suspension.
10. Any concomitant medication for PSP must be well-tolerated and unchanged for at least 1 month prior to Baseline visit and its dose and regimen should be maintained during study if there are no clinical reasons to modify it.
11. Occupational, physical, respiratory, or speech therapy is allowed but it must be stable for at least 1 month prior to screening.
12. Pharmacological treatment of any other chronic condition must be stable and well-tolerated for at least 1 month prior to screening. Analgesics, occasional per request nonsteroidal anti-inflammatory agents, and treatments for transient or emergent conditions are allowed.
13. Signed informed consent by patient and permitted prior to initiation of any study-specific procedure.

Exclusion Criteria:

1. Failure to perform screening or baseline examinations.
2. Hospitalization or change of chronic concomitant medication 1 month prior to or during screening period (apart from pre-planned hospitalization for a condition, which did not deteriorate since 1 month prior to screening period).
3. Clinical, laboratory or neuroimaging findings consistent with:

   * other primary degenerative diseases such as Parkinson's disease; dementia with Lewy bodies; corticobasal degeneration; frontotemporal dementia; multiple system atrophy; parkinsonism-dementia complex of Guam, Kii or Guadeloupe; Alzheimer's disease; amyotrophic lateral sclerosis; Creutzfeldt-Jakob Disease; Huntington's disease; Down's syndrome; etc.
   * cerebrovascular disease as major, strategic or multilacunar infarcts, or extensive white matter lesions scoring 3 in the Wahlund's scale [Wahlund et al., 2001].
   * other central nervous system diseases (hydrocephalus, severe head trauma, tumours, subdural haematoma or other relevant space occupying processes, etc.).
   * epilepsy.
   * other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, clinically significant serum electrolyte disturbances, juvenile onset diabetes mellitus, etc.).
4. A current Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnosis of active major depression, schizophrenia or bipolar disorder.
5. Clinically significant, advanced or unstable disease that may interfere with primary or secondary variable evaluations, may bias clinical or mental assessment or put patient at special risk, such as:

   * chronic liver disease, as indicated by liver function test abnormalities (ALAT, ASAT, bilirubin or GGT out of range) positive serology for Hepatitis C, or other manifestations of liver disease
   * respiratory insufficiency
   * renal insufficiency (serum creatinine >2 mg/dL (>150 micromol/L) and creatinine clearance <60 (according to Cockcroft-Gault formula)
   * heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within 6 months before screening).
   * bradycardia (heart beat <50/min) or tachycardia (heart beat >95/min)
   * episodes of unstable or uncontrolled hypertension (systolic pressure >160 mm Hg or diastolic pressure >100 mm Hg) or hypotension (systolic pressure <90 mm Hg or diastolic pressure <45 mm Hg) during 2 months prior to Baseline visit.
   * atrioventricular block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcF interval (males >450 msec and females >470 msec using Fridericia's formula: QTc = QT/cube root of RR).
   * uncontrolled diabetes mellitus.
   * malignant tumors within last 5 years except skin malignancies (other than melanoma) or indolent prostate cancer.
   * metastases.
6. Disability that may prevent the patient from completing all study requirements (e.g., blindness, deafness, and severe language difficulty).
7. Chronic daily drug intake of:

   * drugs metabolized by cytochrome P450 (CYP)3A4 with narrow therapeutic window (acenocoumarol, warfarin, and digitoxin)
   * anticonvulsants indicated for epileptic seizures
   * systemic anticholinergics with relevant action on central nervous system
   * acetylcholinesterase inhibitors
   * neuroleptics except quetiapine, clozapine or other atypical neuroleptics
   * nootropics such as piracetam, propentofylline, hydergine, vinpocetine, ginkgo biloba, coenzyme Q-10, idebenone and derivatives
   * centrally active anti-hypertensive drugs such as clonidine, alpha methyl dopa, guanidine, and guanfacine
   * systemic cortico-steroids or immunosuppressants
   * systemic nonsteroidal anti-inflammatory agents (except taken as occasional medication per request or acetylsalicylic acid up to 100 mg/day as an antiplatelet agent).
   * memantine, lithium, valproic acid or other GSK-3 inhibitors within 3 months prior to the Baseline visit.
8. Suspected or known history of drug abuse or excessive alcohol intake*
9. Suspected or known allergy to any components of study treatments.
10. Enrollment in another investigational drug study within 3 months before Baseline visit.
11. Any condition, which in the opinion of Investigator makes patient unsuitable for inclusion or likely to be non-compliant.

    * More than 21 units per week for men and 14 for women; or consumption of more than 8 units in a single episode. 1 unit equals approximately 1 glass of wine, 250 ml of beer or 1 shot (25 ml) of spirit.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The change from Baseline between the 2 active study medication groups compared with the placebo group in the Progressive Supranuclear Palsy Rating Scale of Golbe | 52 weeks

SECONDARY OUTCOMES:
Number of AEs and patients with an incidence rate of ≥ 5% AEs | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in Modified Schwab and England Scale | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in Timed Up and Go Test (quantitative motor function) | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in cognitive function(Dementia Rating Scale-2,Frontal Assessment Battery,category and letter verbal fluency) | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in Starkstein Apathy Scale (behavior) | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in functional assessments(Unified Parkinson Disease rating Scale part II and European Quality of Life questionnaire) | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in Clinical Global Impression of Change | 52 weeks
Change from Baseline between 2 active study medication groups vs placebo group in Clinical Global Impression of Severity | 52 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United States (6):
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Department of Neurology, David Geffen School of Medicine at UCLA, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida 5, Tampa, Florida
  - Division of Movement Disorders, University of Louisville, Louisville, Kentucky
  - University of Medicine and Dentistry, Robert Wood Johnson Medical School, New Brunswick, New Jersey
- Germany (6):
  - Neurologisches Fachkrankenhaus für Bewegungsstörungen/Parkinson Beelitz, Beelitz-Heilstätten
  - Humboldt Universitat Charite, Campus Virchow, Neurologisch, Berlin
  - Universitatsklinikum Carl-Guslav-Carus, Technische Universitat Dresden, Klinik und Poliklinik fur Neurologie, Dresden
  - Medizinische Hochschule Hannover, Neurologie 0E 7210, Hanover
  - Zentrum fur Nervenheilkunde. Klinik fur Neurologie mit Poliklinik., Marburg
  - University Hospital Tuebingen,Eberhard-Karls-Universitat, Universitatsklinikum Neurologie, Tübingen
- Spain (9):
  - Fundació Ace, Barcelona, Barcelona
  - Hospital Puerta del Hierro, Madrid, Madrid
  - Hospital de Cruces, Barakaldo
  - Dpto.neurologia. H. Clinic., Barcelona
  - Hospital de Donostia, Donostia / San Sebastian
  - Dpt. Neurologia. Hospital Ramón y Cajal., Madrid
  - Hospital U. La Paz, Madrid
  - Hospital Mutua Terrassa, Terrassa
  - Departement of Neurology, Hospital La Fe, Valencia
- United Kingdom (3):
  - The Walton Centre for Neurology and Neurosurgery NHS Trust, Liverpool
  - Reta Lila Weston Institute of Neurological Studies,Sara Koe PSP Research Centre, London
  - Clinical Ageing Research Unit, Newcastle upon Tyne

REFERENCES:
- [Derived] Hoglinger GU, Schope J, Stamelou M, Kassubek J, Del Ser T, Boxer AL, Wagenpfeil S, Huppertz HJ; AL-108-231 Investigators; Tauros MRI Investigators; Movement Disorder Society-Endorsed PSP Study Group. Longitudinal magnetic resonance imaging in progressive supranuclear palsy: A new combined score for clinical trials. Mov Disord. 2017 Jun;32(6):842-852. doi: 10.1002/mds.26973. Epub 2017 Apr 24. PMID 28436538